CLINICAL TRIAL: NCT01533623
Title: The 1 Year Follow-up of Objective Measures of Oral Appliance Compliance for Treatment of Sleep-disordered Breathing (SDB): a Clinical Trial
Brief Title: The 1 Year Follow-up Objective Oral Appliance Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, principal Investigator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EC 11/41/291
Record Dates: First submitted 2012-01-31; First posted 2012-02-15 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Sleep-disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- mandibular advancement device treatment (Other): Patients diagnosed with sleep-disordered breathing that receive treatment with a titratable, duobloc mandibular advancement devices
  Interventions: Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Mandibular Advancement Device — Nightly wearing time
  Other Names: RespiDent Butterfly® Mandibular Repositioning Appliance

SUMMARY:
The investigators will perform a 1-year clinical trial measuring objective compliance during mandibular advancement device (MAD) treatment.

The investigators will enroll 50 patients that received treatment with a titratable, duobloc MAD (RespiDent Butterfly®, RespiDent, Nijlen, Belgium) and participated in the original study "Objective versus subjective compliance with oral appliance therapy for obstructive sleep apnea hypopnea syndrome", registered at Clinical Trials.gov (NCT01284881).

Active microsensors (TheraMon®,Handelsagentur Gschladt, Hargelsberg, Austria) are provided by the Handelsagentur Gschladt without any costs. The sampling interval of the recording will be done at a rate of 1 measurement per 15 minutes (every 900 seconds). Using this sample interval, the capacity of the active microsensor allows for data acquisition during a 100 day period.

A follow-up appointment is scheduled +/- 265 days after the start of the original study. A second follow-up visit is scheduled again 1 year after the start of the original study.

The objective measurement of MAD wear time (total hours of wear time and the mean hours of wear per night over the respective period) will be based on the assumption that the MAD has been worn when the chip records a temperature intraorally.

DETAILED DESCRIPTION:
This clinical trial is an extension to trial 10/48/340, registered at Clinical Trials.gov (NCT01284881).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of sleep-disordered breathing
* started treatment with a titratable, duobloc mandibular advancement device
* participated in original study 10/48/340 (3 month follow-up of compliance during treatment with mandibular advancement device)

Exclusion Criteria:

* dental exclusion criteria for mandibular advancement devices
* medical contra-indications for mandibular advancement devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of measuring objective mean wearing time | 1 year
  To assess the safety and feasibility of measuring objective mean wearing time as a measure of objective oral appliance wear. The objective mean wearing time will be assessed using a microsensor thermometer. Regular follow-up visits will be performed, and patients will be questioned regarding side-effects of the microsensor.

SECONDARY OUTCOMES:
therapeutic index | 1 year
  to calculate the therapeutic index based on objective compliance and decrease in apnea-hypopnea index / disease severity

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium